CLINICAL TRIAL: NCT03152266
Title: Short-Term Outcome of Surgical Treatment of Osteochondral Impaction in Acetabular Fractures
Brief Title: Function Outcome of Impaction Injuries in Acetabular Fractures
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Bahaaeldin Mohamed Abdelhafez, Principal investigator, Assiut University
Other Study IDs: OCIA
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Acetabular Fracture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention. Observational study — Follow up of the function of the hip after reduction of the impacted fragment which associated with acetabular fractures

SUMMARY:
Is the anatomical reduction of osteochondral impaction in the acetabular fractures will improve the functional outcome? Despite the increasing amount of literature related to the management of anteromedial dome impactions and marginal impactions, there are still remaining issues and controversies pertaining mainly to the exact anatomy and location of the lesion, the best method of reduction, the need and type of subchondral void filling, the best method of stabilization, the need of reduction in elderly population and its true value as an outcome prognostic factor.

DETAILED DESCRIPTION:
The reduction of the impacted fragment done through many ways and techniques , all acetabular approaches can be used to reach to the impacted part or through independent cortical window, The impacted part can be reached through the fracture itself as in marginal impaction through the posterior wall and in anteromedial impaction through the quadrilateral plate. Then using a bone graft as a void filling which can be taken from iliac bone or greater trochanter. Post-operative x-rays and computed tomography scan will be done to all patients , Radiological grading immediate post-operative and at the last follow-up according to Matta , Heterotopic ossification will be classified according to the Brooker classes on an Anteroposterior radiograph, Posttraumatic arthritis will be evaluated according to the method by Kellgren and Lawrence, functional outcome will be assessed according to Merle D'Aubigne and Postel scoring which was modified by Matta, Avascular necrosis of hips will be classified according to Ficat and Arlet classification.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic Osteochondral impaction injuries of the acetabulum (marginal and dome ).
* Pure impaction without cortical interruption
* Closed fractures.
* Skeletally mature (adults and elderly).

Exclusion Criteria:

* Fractures in skeletally immature patients.
* Pathological fractures .
* Associated proximal Hip fractures.
* Open acetabular Fractures.
* Fractures more than 3 weeks

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients will be admitted at emergency department of assiut university hospital , ATLS protocol will be applied , preoperaive plane xray (anteroposterior and CT scan will be done)post operative x rays and CT scan will be done to all patients , Radiological grading just post-operative at the last follow-up according to Matta, Heterotopic ossification was classified according to the Brooker classes on an AP radiograph, Posttraumatic arthritis was evaluated according to the method by Kellgren and Lawrence, functional outcome will be assessed according to Merle d'Aubigne and Postel scoring which was modified by Matta, Avascular necrosis of hips was classified according to Ficat and Arlet classification
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
modified Merle d'Aubigne and Postel scoring | 6th month
  The modified Merle D'Aubigné clinical hip score is the most generally accepted clinical grading system for evaluating the results of acetabular fracture treatment , which evaluates pain, gait and mobility, on a scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martins e Souza P, Giordano V, Goldsztajn F, Siciliano AA, Grizendi JA, Dias MV. Marginal impaction in posterior wall fractures of the acetabulum. AJR Am J Roentgenol. 2015 Apr;204(4):W470-4. doi: 10.2214/AJR.14.12451. PMID 25794097
- [Background] Wu XB, Wang MY, Zhu SW, Cao QY, Wu HH. [Marginal impaction in acetabular fractures]. Zhonghua Wai Ke Za Zhi. 2003 Apr;41(4):289-91. Chinese. PMID 12882675
- [Background] Leucht P, Castillo AB, Bellino MJ. Comparison of tricalcium phosphate cement and cancellous autograft as bone void filler in acetabular fractures with marginal impaction. Injury. 2013 Jul;44(7):969-74. doi: 10.1016/j.injury.2013.04.017. Epub 2013 May 14. PMID 23684351
- [Background] Moed BR, WillsonCarr SE, Watson JT. Results of operative treatment of fractures of the posterior wall of the acetabulum. J Bone Joint Surg Am. 2002 May;84(5):752-8. doi: 10.2106/00004623-200205000-00008. PMID 12004016
- [Background] Bhandari M, Matta J, Ferguson T, Matthys G. Predictors of clinical and radiological outcome in patients with fractures of the acetabulum and concomitant posterior dislocation of the hip. J Bone Joint Surg Br. 2006 Dec;88(12):1618-24. doi: 10.1302/0301-620X.88B12.17309. PMID 17159175
- [Background] Giannoudis PV, Kanakaris NK, Delli Sante E, Morell DJ, Stengel D, Prevezas N. Acetabular fractures with marginal impaction: mid-term results. Bone Joint J. 2013 Feb;95-B(2):230-8. doi: 10.1302/0301-620X.95B2.30548. PMID 23365034
- [Background] Moed BR, Yu PH, Gruson KI. Functional outcomes of acetabular fractures. J Bone Joint Surg Am. 2003 Oct;85(10):1879-83. doi: 10.2106/00004623-200310000-00002. PMID 14563792
- [Background] Ugino FK, Righetti CM, Alves DP, Guimaraes RP, Honda EK, Ono NK. Evaluation of the reliability of the modified Merle d'Aubigne and Postel Method. Acta Ortop Bras. 2012;20(4):213-7. doi: 10.1590/S1413-78522012000400004. PMID 24453605
- [Background] Kreder HJ, Rozen N, Borkhoff CM, Laflamme YG, McKee MD, Schemitsch EH, Stephen DJ. Determinants of functional outcome after simple and complex acetabular fractures involving the posterior wall. J Bone Joint Surg Br. 2006 Jun;88(6):776-82. doi: 10.1302/0301-620X.88B6.17342. PMID 16720773
- [Background] Manson T, Schmidt AH. Acetabular Fractures in the Elderly: A Critical Analysis Review. JBJS Rev. 2016 Oct 4;4(10):e1. doi: 10.2106/JBJS.RVW.15.00090. PMID 27792674
- [Background] Gansslen A, Hildebrand F, Kretek C. Transverse + posterior wall fractures of the acetabulum: epidemiology, operative management and long-term results. Acta Chir Orthop Traumatol Cech. 2013;80(1):27-33. PMID 23452418
- [Background] Giannoudis PV, Tzioupis C, Papathanassopoulos A, Obakponovwe O, Roberts C. Articular step-off and risk of post-traumatic osteoarthritis. Evidence today. Injury. 2010 Oct;41(10):986-95. doi: 10.1016/j.injury.2010.08.003. PMID 20728882
- [Background] Zhuang Y, Lei JL, Wei X, Lu DG, Zhang K. Surgical treatment of acetabulum top compression fracture with sea gull sign. Orthop Surg. 2015 May;7(2):146-54. doi: 10.1111/os.12175. PMID 26033996
- [Background] Bertrand R, Derancourt J, Kassab R. Molecular movements in the actomyosin complex: F-actin-promoted internal cross-linking of the 25- and 20-kDa heavy chain fragments of skeletal myosin subfragment. Biochemistry. 1992 Dec 8;31(48):12219-26. doi: 10.1021/bi00163a035. PMID 1457419
- [Background] Laflamme GY, Hebert-Davies J. Direct reduction technique for superomedial dome impaction in geriatric acetabular fractures. J Orthop Trauma. 2014 Feb;28(2):e39-43. doi: 10.1097/BOT.0b013e318298ef0a. PMID 23681409
- [Background] Tosounidis TH, Stengel D, Giannoudis PV. Anteromedial dome impaction in acetabular fractures: Issues and controversies. Injury. 2016 Aug;47(8):1605-7. doi: 10.1016/j.injury.2016.07.020. No abstract available. PMID 27499274
- [Background] Scolaro JA, Routt ML Jr. Reduction of osteoarticular acetabular dome impaction through an independent iliac cortical window. Injury. 2013 Dec;44(12):1959-64. doi: 10.1016/j.injury.2013.07.012. Epub 2013 Aug 2. No abstract available. PMID 23916899
- [Background] Collinge CA, Lebus GF. Techniques for reduction of the quadrilateral surface and dome impaction when using the anterior intrapelvic (modified Stoppa) approach. J Orthop Trauma. 2015 Feb;29 Suppl 2:S20-4. doi: 10.1097/BOT.0000000000000271. PMID 25486005
- [Background] Jeffcoat DM, Carroll EA, Huber FG, Goldman AT, Miller AN, Lorich DG, Helfet DL. Operative treatment of acetabular fractures in an older population through a limited ilioinguinal approach. J Orthop Trauma. 2012 May;26(5):284-9. doi: 10.1097/BOT.0b013e31821e10a2. PMID 21926638
- [Background] Casstevens C, Archdeacon MT, d'Heurle A, Finnan R. Intrapelvic reduction and buttress screw stabilization of dome impaction of the acetabulum: a technical trick. J Orthop Trauma. 2014 Jun;28(6):e133-7. doi: 10.1097/BOT.0000000000000005. PMID 24296594
- [Background] Lubovsky O, Kreder M, Wright DA, Kiss A, Gallant A, Kreder HJ, Whyne CM. Quantitative measures of damage to subchondral bone are associated with functional outcome following treatment of displaced acetabular fractures. J Orthop Res. 2013 Dec;31(12):1980-5. doi: 10.1002/jor.22458. Epub 2013 Aug 12. PMID 23940014